CLINICAL TRIAL: NCT00546377
Title: A Phase I-II Study of Pentostatin, Cyclophosphamide, Rituximab, and Mitoxantrone in Previously Treated Patients With Chronic Lymphocytic Leukemia and Other Low Grade B-Cell Neoplasms
Brief Title: Pentostatin, Cyclophosphamide, Rituximab, and Mitoxantrone in Treating Patients With Chronic Lymphocytic Leukemia or Other Low-Grade B-Cell Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-077; MSKCC-05077
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; recurrent mantle cell lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; recurrent marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular | interventions — Filgrastim; pegfilgrastim; Rituximab; sargramostim; Cyclophosphamide; Mitoxantrone; Pentostatin; In Situ Hybridization, Fluorescence; Gene Rearrangement; Polymerase Chain Reaction; Flow Cytometry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitoxantrone (Experimental)
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Biological: rituximab; Biological: sargramostim; Drug: cyclophosphamide; Drug: mitoxantrone hydrochloride; Drug: pentostatin; Genetic: fluorescence in situ hybridization; Genetic: gene rearrangement analysis; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Other: flow cytometry; Procedure: biopsy

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Biological: rituximab
Biological: sargramostim
Drug: cyclophosphamide
Drug: mitoxantrone hydrochloride
Drug: pentostatin
Genetic: fluorescence in situ hybridization
Genetic: gene rearrangement analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: flow cytometry
Procedure: biopsy

SUMMARY:
RATIONALE: Pentostatin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving pentostatin together with combination chemotherapy and rituximab may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of mitoxantrone when given together with pentostatin, cyclophosphamide, and rituximab and to see how well it works in treating patients with chronic lymphocytic leukemia or other low-grade B-cell cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of mitoxantrone hydrochloride followed by a phase II study.

* Phase I: Patients receive pentostatin IV, cyclophosphamide IV, and mitoxantrone hydrochloride IV on day 1. Patients also receive rituximab IV on day 1 beginning in course 2. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive pentostatin, cyclophosphamide, rituximab, and mitoxantrone hydrochloride (at the maximum tolerated dose determined in phase I) as in phase I.

All patients receive either pegfilgrastim subcutaneously (SC) on days 1-4 following each course or filgrastim or sargramostim SC beginning 2 days after each course until blood counts recover.

Patients undergo blood collection and bone marrow biopsy periodically for assessment of therapy response by biomarker and laboratory studies. Samples are analyzed for molecular genetics for IgH arrangement by PCR and for response by immunoelectrophoresis. Some samples are analyzed for response by flow cytometry or fluorescence in situ hybridization (FISH).

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 63 patients (18 patients for phase I and 45 patients for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following diseases confirmed by a Memorial Sloan-Kettering Cancer Center (MSKCC) pathologist:

  * Chronic lymphocytic leukemia meeting the following risk criteria as defined by the three-stage Rai system:

    * Intermediate-risk disease meeting the following criteria for active disease as defined by the NCI Working Group:

      * Weight loss
      * Fatigue
      * Fevers
      * Evidence of progressive marrow failure
      * Splenomegaly
      * Progressive lymphadenopathy
      * Progressive lymphocytosis with a rapid doubling time, defined as doubling time less than 6 months and absolute lymphocyte count > 30,000/μL
    * High-risk disease
  * Other low grade B-cell neoplasms, including any of the following:

    * Small lymphocytic lymphoma
    * Follicular lymphoma
    * Waldenstrom macroglobulinemia
    * Marginal zone lymphomas
    * Mantle cell lymphomas
    * Transformed lymphoma
* Previously treated disease

  * Must have received prior cytotoxic therapy
* Malignant lymphocytes must demonstrate B-cells via immunophenotypic or immunohistochemical analysis NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 8 weeks
* Total bilirubin ≤ 2.0 mg/dL (patients with Gilbert disease or autoimmune hemolytic anemia should have an evaluation for other causes of hyperbilirubinemia, but if none are found, may be enrolled regardless of serum bilirubin)
* Total creatinine ≤ 2.0 mg/dL OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Normal cardiac ejection fraction ≥ 50% (increased ejection fraction [at least 5% over rest]) required for study eligibility

  * Borderline (40-50%) ejection fraction must undergo a stress echocardiogram or MUGA scan
* Patients with autoimmune hemolytic anemia or autoimmune thrombocytopenia are eligible for treatment
* Must have undergone consultation with the primary investigator or his/her designee prior to study entry
* No significant active infections
* No ongoing hepatitis B infection, specifically hepatitis B antigen or surface antigen positivity

  * Hepatitis B antibody-positive patients are eligible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* The following concurrent medications are allowed:

  * Intravenous immunoglobulin (IVIG)
  * Erythropoietin, darbepoetin, filgrastim, or sargramostim
  * Cyclosporine (only for patients with cellular immune cytopenias [i.e., pure red cell aplasia]), with required consultation of the principle investigator or designee
* Concurrent prednisone allowed provided it is used as brief courses (≤ 7 days) for inflammatory conditions unrelated to CLL
* No concurrent chemotherapy or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renier Brentjens, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Andrew D. Zelenetz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone: To determine the dose of mitoxantrone that can be safely administered with pentostatin, cyclosphosphamide, and rituximab in previously treated patient with CLL and other low grade B-cell malignancies.
Period: Overall Study
Arm/Group | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone
Started | 50
Completed | 43
Not Completed | 7
Not completed — Deemed ineligible | 1
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Complete response (CR): Absence of lymphadenopathy, hepatomegaly or splenomegaly by physical examination and appropriate radiographic techniques (if abnormal pre-treatment): it is recognized that some patients with lymphoid malignancies who achieve a CR may have mild persistent abnormalities on CT Scan. Such abnormalities if stable on subsequent scanning will not be viewed as persistent disease in patients who otherwise meet the criteria for CR. Response will be assessed on an ongoing basis, but at a minimum of prior to cycle four and following completion of all therapy. Patients who are removed from study early will have response status determined at time of removal from study. The major criteria for determination of response to therapy in patients with CLL include physical examination and examination of the peripheral blood and bone marrow. Radiographic studies are not required but those that were abnormal pre-treatment, will be repeated to document the degree of maximal response.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone
Number analyzed (Participants) | 43
participants
  Complete Response | 11
  Partial Response | 23
  Stable Disease | 4
  Progression of Disease | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Mitoxantrone
Description: The MTD is defined as the highest dose studied for which the incidence of DLT is less than 33%. In the phase I portion of the trial, cohorts of 3-6 pts will receive pentostatin, cyclophosphamide and rituximab along with one of three potential dose levels of mitoxantrone. The following dose escalation scheme will be followed: If none of the initial three pts in a cohort experience a dose-limiting toxicity (grade 4 infection, or grade ≥ 3 non-hematologic toxicity that persists for 7 days or more) then a new cohort of three pts will be treated at the next higher dose level. If one of the three pts in a cohort experiences DLT, then up to three additional pts will be treated at the same dose level. If two or more pts in a cohort experience DLT, then the maximum tolerated dose (MTD) will have been exceeded, and no further dose escalation will occur. The previous dose level will be considered as the MTD.
Time Frame: 2 years
Measure: Number; unit: mg/m2
Arm/Group | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone
Number analyzed (Participants) | 43
mg/m2 | 10

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone
Serious Adverse Events (participants affected / at risk) | 19/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone (N=43)
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 1 (1)
Allerg rhinitis (w sneez, nas stuff, postnas drip) (Immune system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 7 (9)
Fever (in the absence of neutropenia) (General disorders) | 5 (6)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 2 (2)
Infection w/ Gr 3/4 neut, Colon (Infections and infestations) | 1 (1)
Infection w/ Gr 3/4 neut, Sinus (Infections and infestations) | 1 (1)
Infection w/ Gr 3/4 neut, Skin (cellulites) (Infections and infestations) | 1 (1)
Infection, other (Infections and infestations) | 1 (1)
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Pain - Abdomen NOS (Investigations) | 1 (1)
Pain - Head/headache (Investigations) | 2 (3)
Pain - Neck (Investigations) | 1 (1)
Pain - Pelvis (Investigations) | 1 (1)
Pain - Throat/pharynx/larynx (Investigations) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Vasovagal episode (Cardiac disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentostatin,Cyclophosphamide,Rituximab & Mitoxantrone (N=43)
ALT, SGPT (Metabolism and nutrition disorders) | 9 (50)
AST, SGOT (Metabolism and nutrition disorders) | 7 (40)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 (40)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (50)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 9 (20)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (10)
Creatinine (Metabolism and nutrition disorders) | 5 (15)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 31 (50)
Hemoglobin (Metabolism and nutrition disorders) | 31 (100)
INR (Blood and lymphatic system disorders) | 2 (5)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 31 (150)
Lymphopenia (Blood and lymphatic system disorders) | 28 (150)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 31 (150)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 13 (50)
Platelets (Blood and lymphatic system disorders) | 20 (150)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (5)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes